CLINICAL TRIAL: NCT01932229
Title: An Open Label Study of BIBW 2992/Afatinib in Advanced Non-Small Cell Lung Cancer Patients Pre-treated With Erlotinib or Gefitinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-12-9547-JB-CTIL
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: NSCLC
Keywords: Advanced NSCLC; EGFR mutation; TKIs; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Afatinib treatment (Experimental)
  Interventions: Drug: Afatinib treatment

INTERVENTIONS:
Drug: Afatinib treatment

SUMMARY:
Advanced lung cancer (non-small cell lung cancer) with a mutation in the EGFR (epidermal growth factor receptor) gene, which have disease progression after treatment with an EGFR inhibitor (erlotinib or gefitinib), and have progression of disease also after treatment with chemotherapy will be recruited. The trial has only one arm, of afatinib daily treatment. Blood and exhaled breath samples will be collected for investigations aiming to identify factors that predict response to afatinib.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC
* EGFR mutation or six months or longer benefit from EGFR TKIs
* Disease progression on chemotherapy, or inability to receive chemotherapy for medical reasons.
* Disease progression on EGFR TKI, or the presence of an EGFR mutation that does predicts for poor response to first generation EGFR TKIs.

Exclusion Criteria:

* Inability to take oral drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | One year

SECONDARY OUTCOMES:
Overall survival | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gat, Israel